CLINICAL TRIAL: NCT02131701
Title: PPP-Botnia Exercise Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Folkhälsan Researech Center (Other)
Collaborators: Närpes Health Care Center, Närpes, Finland (Unknown); Department of Social Services and Health Care, Jakobstad, Finland (Unknown); Department of Clinical Sciences, Lund University Diabetes Center, CRC, Lund University, Malmö, Sweden (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PPP2007
Record Dates: First submitted 2014-05-04; First posted 2014-05-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Family History of Type 2 Diabetes
Keywords: Physical fitness; Family history of type 2 diabetes; Prescription of exercise
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training group (Active Comparator): The training group received individualized information about moderate training and was also offered training in group twice a week during 12 months. The training included both endurance training (nordic walking, water gymnastics) and training in gym.
  Interventions: Behavioral: Physical activity
- Prescription of exercise (Active Comparator): Individualized sessions for exercise prescription aiming at moderate exercise of 30 minutes at least 5 days a week
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity

SUMMARY:
The aim of the study is to evaluate the long-term effects of a prescription of exercise versus a group-based training program on aerobic fitness, muscle strength and metabolic variables in subjects with poor physical fitness. The participants are further stratified for a family-history of type 2 diabetes. The number of subjects in each group of intervention is planned to be 150, aged 30-70 years and non-diabetic.

Intervention: All study subjects take part in two individual sessions for exercise prescription aiming at moderate exercise of 30 minutes at least 5 days a week. The prescription group perform exercise by themselves, while the training group will be offered supervised physical training, including both endurance training and training in gym twice a week during 12 months.

The subjects will be followed up at 1, 2, 3 and 5 years after the basal visit.

Methods of follow-up: At the study visits physical fitness will be measured by a 2 km walking test, glucose tolerance by oral glucose tolerance test with measurement of glucose and insulin. Lipids will be measured. Questionnaires will be used to follow lifestyle, physical activity, cardiovascular disease and medication.

In the training group 30 subjects with and 30 subjects without a family history of type 2 diabetes will participate in a sub-study including muscle- and fat-biopsy before the start of the study, after 1 and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* poor physical fitness based on repeated walking test (UKK 2 km walking test)
* non-diabetic

Exclusion Criteria:

* health problems complicating moderate physical training

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2006-10; Primary Completion 2008-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
improvement in physical fitness | will be measured at 1, 2,3 and 5 years
  Fitness will be measured by a 2 km walking test, which is an indirect measure of oxygen uptake

SECONDARY OUTCOMES:
changes in body composition | measured at 1, 2, 3 and 5 years
  body composition will be measured as weight, waist, fat percentage

OTHER OUTCOMES:
changes in muscle strength | will be measured before study and after 1 and 5 years
  muscle strength will be followed by the method of one repetition maximum

CONTACTS AND LOCATIONS:
Overall Officials: Bo Isomaa, MD, Principal Investigator — Folkhälsan Research Center, Helsinki, Finland
Locations (1):
- Folkhälsan Research Center, Helsinki, Finland

REFERENCES:
- [Derived] Wasenius NS, Isomaa BA, Ostman B, Soderstrom J, Forsen B, Lahti K, Hakaste L, Eriksson JG, Groop L, Hansson O, Tuomi T. Low-cost exercise interventions improve long-term cardiometabolic health independently of a family history of type 2 diabetes: a randomized parallel group trial. BMJ Open Diabetes Res Care. 2020 Nov;8(2):e001377. doi: 10.1136/bmjdrc-2020-001377. PMID 33219117